CLINICAL TRIAL: NCT00525447
Title: A Phase I Study of SGN-40 (Anti-huCD40 mAb), Lenalidomide (Revlimid®, cc 5013), and Dexamethasone in Patients With Multiple Myeloma (MM)
Brief Title: Study of SGN-40, Lenalidomide, and Dexamethasone in Patients With Multiple Myeloma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Seagen Inc. (Industry)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SG040-0006
Record Dates: First submitted 2007-08-31; First posted 2007-09-05 (Estimated); Last update posted 2014-10-09 (Estimated); Status verified 2014-10

CONDITIONS: Multiple Myeloma
Keywords: Antigens, CD40; Antibodies, Monoclonal; Combined Modality Therapy; Multiple Myeloma; Blood Coagulation Disorders; Hematologic Diseases; Hemorrhagic Disorders; Hemostatic Disorders; Immunoproliferative Disorders; Lymphoproliferative Disorders; Paraproteinemias; Vascular Diseases; Antibody-Dependent Cell Cytotoxicity
MeSH Terms: conditions — Multiple Myeloma; Blood Coagulation Disorders; Hematologic Diseases; Hemorrhagic Disorders; Hemostatic Disorders; Immunoproliferative Disorders; Lymphoproliferative Disorders; Paraproteinemias; Vascular Diseases | interventions — dacetuzumab; Lenalidomide; Dexamethasone; Calcium Dobesilate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: SGN-40; Drug: lenalidomide; Drug: dexamethasone

INTERVENTIONS:
Drug: SGN-40 — 2-12 mg/kg IV (in the vein) on Days 1, 4, 8, 15, and 22 of Cycle 1; 4-12 mg/kg IV (in the vein) on Days 1, 8, 15, and 22 of Cycles 2-4; 4-12 mg/kg IV (in the vein) on Days 1, 8, and 15 of Cycles 5-8.
  Other Names: dacetuzumab
Drug: lenalidomide — Up to 25 mg daily of a 21-day cycle.
  Other Names: Revlimid
Drug: dexamethasone — 40 mg administered weekly.
  Other Names: Decadron

SUMMARY:
This is a Phase I, open-label, multi-dose trial to define the MTD and tolerability of a regimen including lenalidomide, dexamethasone, and intravenous SGN-40 in patients with relapsed multiple myeloma.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of multiple myeloma.
* Received at least one prior systemic therapy other than single-agent corticosteroids.
* Measurable disease of monoclonal protein greater than or equal to 0.5 gram/dL in plasma or 0.5 gram/24 hr urine collection, or greater than 10 mg/dL free light chain (FLC) in serum as determined by serum FLC assay and provided the serum FLC ratio is abnormal.

Exclusion Criteria:

* Received an allogenic stem cell transplant.
* Previous intolerance of lenalidomide or dexamethasone.
* Primary invasive malignancy (other than multiple myeloma) within the last 3 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2007-08; Primary Completion 2010-01 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Adverse events and lab abnormalities. | Within 3 weeks of final infusion of SGN-40

SECONDARY OUTCOMES:
Best clinical response, progression-free survival, and overall survival. | Study duration
PK profile. | Within 3 weeks of final infusion of SGN-40
Anti-drug antibody immune responses. | Within 3 weeks of final infusion of SGN-40

CONTACTS AND LOCATIONS:
Overall Officials: Nancy Whiting, PharmD, Study Director — Seagen Inc.
Locations (9):
- United States (9):
  - Rocky Mountain Cancer Center, Denver, Colorado
  - H. Lee Moffitt Cancer Center & Research Institute, Tampa, Florida
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Weill Medical College of Cornell University, New York, New York
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Baylor University Medical Center, Dallas, Texas